CLINICAL TRIAL: NCT04809805
Title: An Open Label, Phase 1, First-in-human, Study to Evaluate Safety, Tolerability, Maximum Tolerated or Administered Dose, Pharmacokinetics, Pharmacodynamics and Tumor Response Profile of Schlafen12 Complex Inducer (SLFN12 ci) BAY 2666605 in Participants With Metastatic Melanoma and Other Advanced Solid Tumors.
Brief Title: A Study to Learn How Safe BAY2666605 is, How it Affects the Body, How it Moves Into, Through and Out of the Body, the Maximum Amount That Can be Given and Its Action Against Tumors in Adult Participants With Skin Cancer That Has Spread to Other Parts of the Body and Other Types of Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the high probability of not achieving a therapeutic window and lack of evidence of sufficient clinical benefit.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 20733
Record Dates: First submitted 2021-03-05; First posted 2021-03-22 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Melanoma and Other Solid Tumors
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation of BAY2666605 (Experimental): Approximately 7 or 8 dose levels are planned.
  Interventions: Drug: BAY2666605
- Dose expansion of BAY2666605 (Experimental): Participants will receive BAY 2666605 at the dose and regimen declared safe in the dose escalation part.
  Interventions: Drug: BAY2666605

INTERVENTIONS:
Drug: BAY2666605 — One oral solution strength of BAY2666605 will be used. Two different tablet strengths of BAY2666605 will be available.

SUMMARY:
Researchers are looking for a better way to treat people who have advanced cancer.

In this study researchers want to learn more about a new substance called BAY2666605. BAY2666605 triggers the formation of a complex of two proteins called SLFN12 and PDE3A. This complex drive cancer cells into cell death by a mechanism called apoptosis. The complex is only formed in the cancers which contain both proteins.

This study is done in adult patients who have certain types of advanced cancers that cannot be cured by drugs that are currently available. The cancer types include skin cancer that has spread to other parts of the body and cancer that started in the bones or soft tissue, the ovaries, or the brain. Patients with these cancers are only included if the cells of the patient's cancer contain the building plan to produce SLFN12-phosphodiesterase 3A (PDE3A) complex. To confirm this, a specific test is performed with the cancer cells.

The researchers will study how BAY2666605 moves into, through and out of the body. Researchers will try to find the best dose that can be given, how safe BAY2666605 is and how it affects the body. Researchers will also study the action of BAY2666605 against the cancer. Part A will include about 36 participants and up to another 12 participants. Part B will include about 41 participants. All of the participants will take BAY2666605 by mouth as either a liquid or as tablets.

During the study, the participants will take the treatment in 4 week periods called cycles. In each cycle, the participants will in general take BAY2666605 once daily. The participants may also be asked to do overnight fasting before the intake of substance and to have standard high-fat, high-calorie breakfast on some days before taking the dose.

These 4 week cycles will be repeated throughout the trial. The participants can take BAY2666605 until their cancer gets worse, until they have medical problems, or until they leave the trial. Participants will have around 18 visits in each cycle. Some of the visits can also be done via Phone.

During the trial, the study team will take blood and urine samples, do physical examinations and check the participants' heart health using an electrocardiogram (ECG) and an ultrasound of the heart. The study team will also take pictures of the participants' tumors using CT or MRI scans. The study team will ask how the participants are feeling, if participants have any medical problems or if participants are taking any other medicine. About 1 month and 3 months after the last dose, the participants will have another visit and a phone call respectively where participants will be checked for and asked about medical problems. The researchers will then contact the participants every 3 months until the trial ends.

ELIGIBILITY:
Inclusion Criteria:

Pre-screening:

* Signed informed consent for pre-screening
* Male or female participants aged ≥ 18 years
* Participants with histologically confirmed diagnosis of melanoma, glioblastoma/anaplastic astrocytoma, sarcoma or epithelial ovarian cancer/fallopian tube/primary peritoneal cancer
* Availability of archival tumor tissue (5-10 for prescreening, further 20 to be provided at screening)
* ECOG ≤2

Main Screening :

* Positive SLFN12/PDE3A expression in archival tumour
* Minimum life expectancy at least 12 weeks
* Documented radiological disease progression after treatment with all available standard of care therapies for advanced/metastatic disease and at least one measurable lesion
* Adequate bone marrow, liver, and renal function
* Adequate blood clotting
* Left ventricular ejection fraction >50%
* All AEs due to previous therapies to CTCAE Grade ≤1. Grade ≤2 neuropathy, fatigue, alopecia, or anorexia, for which further resolution is not expected, may be eligible.
* Negative pregnancy test and use of highly effective contraception
* Signed informed consent for main screening

Exclusion Criteria:

Pre-screening:

* Any malabsorption conditions
* Known HIV infection, active HBV or HCV infection
* Known hypersensitivity to PDE3 inhibitors, or excipients in the formulation; concomitant treatment with any other PDE3 inhibitors
* Participants with clinically relevant cardiovascular diseases and/or relevant ECG findings
* Participants with history of hemorrhage, bleeding disorders or platelet function abnormalities, aneurysm or aneurysmal vasculopathy; Participants with arterial thromboembolic events (ATEs) or venous thromboembolic events (VTEs), including transient ischemic attacks or pulmonary embolism within 6 months before the start of BAY 2666605 or deep vein thrombosis within 3 months before the start of BAY 2666605; Participant with a history of gastrointestinal (GI) ulcerations or perforation, fistula formation involving any internal organs.

Main screening

* Moderate or severe hepatic impairment
* History of organ allograft transplantation, including allogeneic bone marrow
* Previous of co-existing cancer(s) distinct in primary site or histology from the cancer evaluated in this study (with few exceptions)
* Participants with any history of primary meningeal tumors and/or Any active symptomatic or untreated central nervous system (CNS) metastases and/or a number of prior and concomitant therapies
* Major surgery, significant trauma, serious non-healing wound, wound healing complications, ulcer or bone fracture within 4wks prior to 1st dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of TEAEs including TESAEs | Up to 6 months after the last participant's first study intervention or until the end of the study, whichever comes first.
  TEAEs: Treatment emergent adverse events; TESAEs:Treatment emergent serious adverse events
The incidence of DLTs at each dose level in the Dose Escalation part of the study | Up to 28 + 14 days
  DLT: Dose limiting toxicity
Maximal plasma exposure (Cmax) of BAY2666605 | Cycle 1 Day 1
AUC(0-24) of BAY2666605 | Cycle 1, Day 1
RP2D of BAY2666605 | Up to 6 months after the last participant's first study intervention or until the end of the study, whichever comes first.
  RP2D: Recommended phase 2 dose. RP2D will be defined in the expansion part.
Cmax,md of BAY2666605 | Cycle 1, Day 15
AUC(0-24)md of BAY2666605 | Cycle 1, Day 15

SECONDARY OUTCOMES:
ORR | Up to 6 months after the last participant's first study intervention or until the end of the study, whichever comes first.
  ORR: Objective response rate
DCR | Up to 6 months after the last participant's first study intervention or until the end of the study, whichever comes first.
  DCR: Disease control rate
DOR | Up to 6 months after the last participant's first study intervention or until the end of the study, whichever comes first.
  DOR: Duration of response
PFS by investigator assessment | Up to 6 months after the last participant's first study intervention or until the end of the study, whichever comes first.
  PFS: Progression-free survival
OS | Up to 6 months after the last participant's first study intervention or until the end of the study, whichever comes first.
  OS: Overall survival

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Sarah Cannon Development Innovations, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics | START San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/20733